CLINICAL TRIAL: NCT00323583
Title: Phase II Study of Paclitaxel, Oxaliplatin, Leucovorin and 5-Fluorouracil (POLF) in Gemcitabine-Refractory Advanced Pancreatic Cancer
Brief Title: Weekly Dosing of an Integrative Chemotherapy Combination to Treat Advanced Pancreatic Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seattle Cancer Treatment and Wellness Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTCA06-02
Record Dates: First submitted 2006-05-05; First posted 2006-05-09 (Estimated); Last update posted 2007-05-08 (Estimated); Status verified 2007-05

CONDITIONS: Adenocarincoma of Pancreas; Stage III Pancreatic Cancer; Stage IVA Pancreatic Cancer; Stage IVB Pancreatic Cancer
Keywords: Cancer; Pancreatic Cancer; Cancer Alternative Therapies; Living with Cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasms | interventions — Paclitaxel; Oxaliplatin; Leucovorin; Fluorouracil; Glutathione; Calcium; Magnesium; Drug Therapy; Complementary Therapies

INTERVENTIONS:
Drug: paclitaxel
Drug: oxaliplatin
Drug: leucovorin
Drug: 5-fluorouracil
Drug: glutathione
Drug: calcium and magnesium
Procedure: Chemotherapy
Procedure: Chemoprotection
Procedure: Complementary and alternative therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as paclitaxel, oxaliplatin, leucovorin and 5-fluoruracil, work in different ways separately and in combination to stop tumor cells from dividing so they stop growing or die. The use of metronomic dosing of chemotherapy minimizes side effects and increases efficacy by anti-angiogenic effects. The pilot study demonstrated promising responses in all patients. It is not yet known how effective this drug and dosing combination is in treating advanced pancreatic cancer.

PURPOSE: This non-randomized phase II trial is studying giving weekly doses of paclitaxel, oxaliplatin, leucovorin and 5-fluorouracil together as second or third-line therapy in treating patient with locally advanced unresectable or metastatic adenocarcinoma of the pancreas following demonstrated progression after first-line gemcitabine.

DETAILED DESCRIPTION:
OBJECTIVES:

* The primary objective is to determine the effectiveness the chemotherapy combination in improving the experience of those with advanced pancreatic cancer in

  * Pain control and other aspects of quality of life
  * Reduction of the tumor size or stabilization of tumor growth
  * Progression free survival
  * Overall survival
* The secondary objective is to determine the safety of this chemotherapy combination by monitoring and the managing the potential side effects

DOSE REGIMEN OUTLINE: Paclitaxel 60mg/m2 IV weekly; Oxaliplatin 50mg/m2 IV weekly; Leucovorin 20 mg/m2 IV weekly, minimum of 40 mg; 5FU 425mg/m2 IV weekly; Weekly for 12 weeks; Calcium and magnesium 1gram each IV prior to and after Oxaliplatin therapy; Glutathione 1500mg/m2 prior to Oxaliplatin

DURATION OF STUDY PERIOD: Patient will continue study treatment until death, disease progression, unacceptable toxicity, patient refusal, or treatment delay greater than 3 weeks, 12 weeks initially, can than continue at discretion of investigator.

EXPECTED NUMBER OF PATIENTS: A total of 80 patients (40 second line of treatment and 40 third line or greater of treatment) will be enrolled for this study beginning in May 2006.

QUALITY OF LIFE: Quality of life will be assessed at baseline, each month of treatment and at the end of study therapy.

ELIGIBILITY:
DISEASE CHARACTERISTICS

Patients with pathologically-proven pancreatic adenocarcinoma, who

1. are not candidate for surgery
2. are not candidate for radiation therapy and
3. have failed gemcitabine-based chemotherapy regimen

Gender Eligible for Study:

* Both

Prior Therapy:

* For advanced disease allowed as above;
* Oxaliplatin or 5-FU will be allowed but a subset analysis will be done for this group of patients;
* Tarceva and/or Erbitux allowed, but subset analysis will be done.

Allergies:

* No known allergy to one of the study drugs

PATIENT CHARACTERISTICS:

* No CNS metastases
* No peripheral neuropathy > grade 2
* ECOG Performance Status <=2
* Age ≤ 65
* No other serious concomitant illness
* Fully recovered from any prior therapy

Lower Age Limit:

* >18

Upper Age Limit:

* ≤ 65

Laboratory:

* ANC >1500
* Platelets >75,000
* Creatinine <=2.0

Other:

* For female patient of childbearing potential, neither pregnant nor breastfeeding, and under active contraception

Exclusion Criteria:

* Performance state >=3
* Uncontrolled serious concomitant disease
* Radiotherapy within the 6 weeks before Cycle 1' Day 1
* Surgery within the 2 weeks before Cycle 1' Day 1

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2006-05

PRIMARY OUTCOMES:
Clinical response rate (PS improvement by ECOG score, analgesic dose reduction)
Response Rate Recist (Uni-Dimensional) Criteria
Progression free survival
Median survival
Overall survival
Quality of life

SECONDARY OUTCOMES:
Tolerance and Safety NCI-CTC version 2

CONTACTS AND LOCATIONS:
Overall Officials: Ben Chue, MD, Principal Investigator — Seattle Cancer Treatment and Wellness Center
Locations (1):
- Seattle Cancer Treatment and Wellness Center, Seattle, Washington, United States